CLINICAL TRIAL: NCT05393440
Title: A First-in-human Phase I Two-stage Clinical Trial for Intratumoral Injection of Recombinant Oncolytic Type II Herpes Simplex Virus (BS-006) in Patients With Recurrent Cervical Cancer
Brief Title: First-in-human (FIH) Phase I Trial of BS-006 in Cervical Cancer
Acronym: CC-OV01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Collaborators: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hui Qiu, Chief Physician and Director of Department of Radiation and Clinical Oncology (Gynaecological Oncology, Wuhan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CC-OV01
Record Dates: First submitted 2022-05-19; First posted 2022-05-26 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Uterine Cervical Neoplasms; Oncolytic viruses; BS-006; Phase I clinical trial; Investigator initiated trial
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-escalation cohort (Experimental): Three subjects will be enrolled in this cohort. First subject will receive first injection in dose level of 1 million CCID50/mL. If tolerated, second injection for this subject will be accelerated to 10 millions CCID50/mL. If tolerated, the third injection will be further accelerated to 100 million CCID50/mL. The maximum volume for per injection time point is 8 mL. Injection will repeat every two weeks until disease progression or unacceptable toxicity or withdrawn of consent or no lesion suitable for injection or death. If dose limiting toxicity (DLT) happens in any dose level, the injection dose will be decrease to the last tolerable level.
  Interventions: Biological: BS-006
- Dose-expansion cohort (Experimental): Fifteen subjects will be enrolled in this cohort. The maximal tolerable dose (MTD) confirmed in the first stage will be utilized in 15 patients. This stage should not be initiated before the completion of dose escalation of all three subjects in the first stage. Treatment will be repeated every two weeks until disease progression or unacceptable toxicity or withdrawn of consent or no lesion suitable for injection or death. Dose interruption, not reduction, is permitted. Treatment will be terminated if toxicity-related treatment interrupt is longer than 28 days. Radiology assessment will be conducted every six weeks.
  Interventions: Biological: BS-006

INTERVENTIONS:
Biological: BS-006 — BS-006 is an engineered recombinant type II herpes simplex virus (HSV2) designed and produced by Wuhan Binhui Biopharmaceutical Co., Ltd. It was derived from HSV2 strain HG52. ICP34.5 and ICP47 genes were deleted to ensure abortive infection and immune destruction in normal cells. Bispecific T cell engager of anti-CD3 antibody and anti-PD-L1 antibody were constructed and inserted into HG52 strain genome.
  Other Names: Recombinant oncolytic type II herpes simplex virus

SUMMARY:
This is a two-stage phase I clinical trial with oncolytic viruses BS-006 in recurrent or metastasis cervical cancer patients who failed in second line treatment.

DETAILED DESCRIPTION:
This trial includes accelerated dose-escalation stage and dose-expansion stage. An engineered modification oncolytic viruses, BS-006, derived from type II herpes simplex virus strain are planed to be injected into the tumor every two weeks until disease progression or unacceptable toxicity or withdrawn of consent or no lesion suitable for injection or death. In dose-escalation stage, there are three dose levels (1 million, 10 millions, 100 millions 50 % cell culture infectious dose (CCID50)/ml) . Treatment dose will escalate to next higher level if no dose limiting toxicity happens for one time of injection in 3 subjects. Maximal tolerable dose is defined as the highest dose with no more than one dose limiting toxicity and is recommended for dose expansion stage. In dose-expansion stage, 15 subjects will be enrolled. BS-006 viruses will be injected into proper tumor lesions every 2 weeks until disease progression or unacceptable toxicity or withdrawn of consent or no lesion suitable for injection or death. Radiology assessment will repeat every 6 weeks. Dose interruption, not reduction, is permitted in this stage.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old and younger than 75 years old;
2. Zubrod-ECOG-WHO performance status is 0-1;
3. Life expectancy is longer than 3 months;
4. Pathologically proven malignant tumor originating from cervix uterine. All pathological types are acceptable except for sarcoma of any subtypes;
5. Radiological confirmed progression after at least 2 lines prior treatment or intolerable toxicity events occur during the second or later line treatment: 1) Neoadjuvant or adjuvant chemotherapy for no less than 2 cycles should be regarded as a separate treatment line if disease progress within 6 months after treatment finish;2) Regional treatment such as brachytherapy, radiofrequency ablation and artery embolization therapy should not be considered as a treatment line; 3) Treatment shift due to toxicity without radiological progression should not be counted as a separate line;
6. At least one measurement lesion according to RECIST 1.1;
7. At least one lesion with maximum diameter is larger than 1cm and surgically accessibility;
8. Patients must have recovered from prior treatment related toxicity to CTCAE grade 1 or 0;
9. Time interval to last systematic treatment or radiation affecting more than 20% bone marrow must be more than 4 weeks;
10. Time interval to last major surgery must be more than 4 weeks;
11. Abundant organ function: 1) Absolute neutrophil count is more than 1500/mm3 without granulocyte colony stimulating factor in the prior 7 days or long-acting granulocyte colony stimulating factor in the prior 20 days; platelets count is more than 100,000/mm3 without thrombopoietic drugs in the prior 7 days or platelet transfusion in the prior 10 days; hemoglobin is more than 9.0g/dL without red blood cell transfusion in the prior 20 days; 2) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are lower than 2.5-fold upper limit of normal (ULN); serum bilirubin is lower than 1.5-fold ULN; serum albumin is more than 3g/dL; 3) Serum creatinine is lower than 1.5-fold ULN; 4) Prothrombin time and activated partial thromboplastin time is lower than 1.3-fold ULN;
12. Patients must have fully recovered from suspected or diagnosed genital herpes beyond 3 months;
13. Patients or their legally authorized representative must be willing and able to sign the informed consent form (ICF) and to adhere to the protocol requirement;
14. Women of childbearing potential must agree to use highly effective contraceptive methods in while on study drug and for at least 3 months after the last injection of BS-006. The pregnancy test within 7 days prior to the first injection must be negative.

Exclusion Criteria:

1. Cervical sarcoma of any subtype or prior history of other malignancy within 5 years;
2. Central nerve system metastasis;
3. Lesions met the requirement outlined in the inclusion criteria are unsafe for injection evaluated by investigators;
4. Severe comorbidities of any organs, including but not limit to myocardial infarction within 6 months, unstable angina pectoris, congestive heart failure, grade 3 or higher hypertension per CTCAE, cardiac arrhythmias, uncontrolled diabetes, fever of unknown reason, active digest ulcer and chronic obstructive pulmonary disease;
5. History of central nervous system infectious or demyelinating disease;
6. Severe infectious disease requiring constant antibiotic treatment;
7. Systematic glucocorticoids use within 2 weeks or glucocorticoids need for a long term;
8. Active infection of hepatitis B or C, HIV, cytomegalovirus, syphilis or other virus requiring treatment;
9. Immune disorder disease;
10. Antiviral treatment of any kinds;
11. Prior participant in experimental viral therapy;
12. Allergy to herpes simplex virus vaccine;
13. Participation in another research study within 4 weeks;
14. Poor compliance or incapacitated patients due to mental illness or other reasons;
15. Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerable dose | 2 months after initiation of enrollment
  The dose level at which there is no more than one DLT happens in dose-escalation stage
Rate and grade of adverse events | From enrollment to 90 days after last treatment of all subjects
  The incidence of adverse events and severity graded according to CTCAE 5.0
Cope numbers of BS-006 | 1 hours predose and 0.5 hours post-dose for first three doses and 1 hours predose ever after
  Detection of BS-006 virus copy numbers in urine, stool, saliva, blood and wiper of injection point and perineum

SECONDARY OUTCOMES:
Tumor response rate | Up to 2 years
  Tumor change assessed by investigator according to RECIST 1.1
Abscopal effect rate | Up to 2 years
  Rate of subjects who showed tumor shrinkage for any untreated lesion
Progression free survival rate | Up to 2 years
  Proportion of participants without tumor recurrence or death
Overall survival rate | Up to 2 years
  Proportion of survival participants

CONTACTS AND LOCATIONS:
Overall Officials: Hui Qiu, Ph. D., Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mondal M, Guo J, He P, Zhou D. Recent advances of oncolytic virus in cancer therapy. Hum Vaccin Immunother. 2020 Oct 2;16(10):2389-2402. doi: 10.1080/21645515.2020.1723363. Epub 2020 Feb 20. PMID 32078405
- [Background] Kohlhapp FJ, Kaufman HL. Molecular Pathways: Mechanism of Action for Talimogene Laherparepvec, a New Oncolytic Virus Immunotherapy. Clin Cancer Res. 2016 Mar 1;22(5):1048-54. doi: 10.1158/1078-0432.CCR-15-2667. Epub 2015 Dec 30. PMID 26719429
- [Background] Andtbacka RH, Kaufman HL, Collichio F, Amatruda T, Senzer N, Chesney J, Delman KA, Spitler LE, Puzanov I, Agarwala SS, Milhem M, Cranmer L, Curti B, Lewis K, Ross M, Guthrie T, Linette GP, Daniels GA, Harrington K, Middleton MR, Miller WH Jr, Zager JS, Ye Y, Yao B, Li A, Doleman S, VanderWalde A, Gansert J, Coffin RS. Talimogene Laherparepvec Improves Durable Response Rate in Patients With Advanced Melanoma. J Clin Oncol. 2015 Sep 1;33(25):2780-8. doi: 10.1200/JCO.2014.58.3377. Epub 2015 May 26. PMID 26014293
- [Background] Raja J, Ludwig JM, Gettinger SN, Schalper KA, Kim HS. Oncolytic virus immunotherapy: future prospects for oncology. J Immunother Cancer. 2018 Dec 4;6(1):140. doi: 10.1186/s40425-018-0458-z. PMID 30514385